CLINICAL TRIAL: NCT03510052
Title: Diet Modification Program for Senior Women With Fecal Incontinence
Brief Title: Diet and Fecal Incontinence in Senior Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 825518
Record Dates: First submitted 2018-04-06; First posted 2018-04-27 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Accidental Bowel Leakage; Fecal Incontinence; Incontinence; Bowel Incontinence
Keywords: diet; Fecal Incontinence; FI; ABL
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet Modification Pilot Program (Other): Investigator will administer DMP which will include a review of the booklets and any targeted recommendations based on the participant's food and symptom diary. The participant will follow the DMP for 6 weeks and report for a follow-up visit.
  Interventions: Behavioral: Diet Modification Pilot Program (DPM)

INTERVENTIONS:
Behavioral: Diet Modification Pilot Program (DPM) — Investigator will administer DMP which will include a review of the booklets and any targeted recommendations based on the participant's food and symptom diary. The participant will follow the DMP for 6 weeks and report for a follow-up visit.

SUMMARY:
Investigators will conduct a single-arm pre-post intervention pilot study in 46 older women with Fecal Incontinence (FI), also known as Accidental Bowel Leakage (ABL). FI symptoms and stool metabolites will be measured at baseline. Intervention with the Diet Modification Program (DMP) will be administered. FI symptoms and stool metabolites will be measured after 6weeks of the intervention.

DETAILED DESCRIPTION:
Study Procedure: Visit Schedule

Visit 1(Baseline visit): Following consent, the study coordinator will obtain participant's demographic data including age, race/ethnicity, body mass index. Data on medical comorbidities, surgical history and medications known to be associated with FI will be collected. The participant's severity of FI will be measured using the St. Mark's Vaizey scale (Vaizey). The impact of FI on quality of life will be measured using the Fecal Incontinence Quality of Life scale (FIQL). The presence, type, and severity of other pelvic floor symptoms known to be associated with FI will be assessed using the Pelvic floor Distress Inventory- Short Form. Participants will be given a Food and Bowel Symptom diary and a stool collection kit at the conclusion of the visit.

Visit 2(Intervention visit): Stool sample will be collected by the study coordinator. Investigators will administer the DMP. Participants will be given the booklet outlining the DMP and investigators will review the participant's Food and Symptom diary and provide targeted recommendations. The participant will be given a second Food and Symptom diary and stool collection kit to return 6 weeks after the intervention start date.

Calls: Trained Nutritionists will call the participant between weeks 2 and 4 for three unannounced 24h diet recall. The 24-hour dietary recalls will be collected using Nutrition Data System for Research, a computer-based software application that facilitates the collection of recalls in a standardized fashion.

Visit 3 (Follow up visit): Post intervention stool samples and Food and Symptom diary will be collected. Questionnaires including the Vaizey, FIQL, Pelvic Floow Disability Index (PFDI), and Patient Global Index of Improvement (PGI-I) will be administered by the study coordinator. Participants will receive compensation for participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years,
2. FI defined as any uncontrolled loss of liquid or solid fecal material that occurs at least monthly over the last 3 months that is bothersome enough to desire treatment,
3. adequate mobility for independent toileting,
4. ability for independent completion of food symptom diary,
5. has some control of her diet and is able to make adjustments
6. able to read and communicate in English,
7. willing to give informed consent

Exclusion Criteria:

1. Currently receiving another treatment for FI
2. significant cognitive impairment at baseline
3. residence in a care facility that provides meals (participants who are not able to adjust their diet will be excluded because the intervention focuses on the participant, not their care facility)
4. current bloody diarrhea,
5. current or past diagnosis of colorectal

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in FI Symptoms (Vaizey) | 6 weeks
  Changes in the participant's symptom severity will be assessed from baseline to study conclusion.

OTHER OUTCOMES:
Changes in stool metabolites | 6 weeks
  Change from baseline in levels of stool deoxycholic acid(DCA, µmol/g feces)

CONTACTS AND LOCATIONS:
Overall Officials: Uduak U Andy, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States